CLINICAL TRIAL: NCT06780449
Title: Long-term Efficacy and Safety of Cagrilintide s.c. 2.4 mg in Combination With Semaglutide s.c. 2.4 mg (CagriSema 2.4 mg/2.4 mg) Once Weekly Versus Placebo in Participants With Obesity
Brief Title: A Research Study to Look Into the Long-term Effect on Weight Loss of CagriSema in People With Obesity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-7859; U1111-1304-7430 (Other: World Health Organization (WHO)); 2024-512144-39 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) after a dose escalation period of 16 weeks during the maintenance period for 88 weeks in the main phase. Participants randomised to this arm will be included in the extension phase for one year.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide and semaglutide subcutaneously once weekly for 104 weeks. Participants randomised to this arm will be included in the extension phase for one year.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive cagrilintide subcutaneously.
  Arms: CagriSema
Drug: Semaglutide — Participants will receive semaglutide subcutaneously.
  Arms: CagriSema
Drug: Placebo cagrilintide — Participants will receive placebo matched to cagrilintide subcutaneously.
  Arms: Placebo
Drug: Placebo semaglutide — Participants will receive placebo matched to semaglutide subcutaneously.
  Arms: Placebo

SUMMARY:
This study will look at how well CagriSema helps people with obesity lose weight compared to a "dummy medicine". CagriSema is a new medicine developed by Novo Nordisk. CagriSema cannot yet be prescribed by doctors. The study has two parts: First part is called the main phase and will last for 2 years, and second part is called the extension phase and will last for 1 year. In the main phase participants will either get CagriSema or "dummy medicine". Which treatment participants get is decided by chance and is not known by participants or the study doctor. In the extension phase participants will get either CagriSema or slowly reduce participants dose of CagriSema if participants had CagriSema in the main phase. Which treatment participants get is decided by chance and is not known by participants or the study doctor in both phases. If participants had "dummy medicine" in the main phase, participants will get CagriSema in the extension phase. Like all medicines, the study medicine may have side effects.

ELIGIBILITY:
Inclusion criteria:

* Male or female.
* Age above or equal to 18 years at the time of signing informed consent.
* Body mass index (BMI) greater than or equal to (>=) 35.0 kilograms per meter square (kg/m^2).

Exclusion criteria:

* Glycated haemoglobin (HbA1c) >= 6.5 percent (48 millimoles per mole [mmol/mol]) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2028-08-28 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to week 104
  Measured in percentage (%).

SECONDARY OUTCOMES:
Number of participants who achieve greater than or equal to (>=) 20 percent body weight reduction | From baseline (week 0) to week 104
  Measured as count of participants.
Number of participants who achieve >= 25 percent body weight reduction | From baseline (week 0) to week 104
  Measured as count of participants.
Number of participants who achieve >= 30 percent body weight reduction | From baseline (week 0) to week 104
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to week 104
  Measured in centimeter (cm).
Change in waist to height ratio | From baseline (week 0) to week 104
  Measured as ratio.
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to week 104
  Measured in millimeter of mercury (mmHg).
Ratio to Baseline in Lipids: Total Cholesterol | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: High Density Lipoprotein (HDL) Cholesterol | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: Low Density Lipoprotein (LDL) Cholesterol | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: Very Low Density Lipoprotein (VLDL) Cholesterol | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: Triglycerides | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: Free fatty acids | From baseline (week 0) to week 104
  Measured as ratio.
Ratio to Baseline in Lipids: Non-HDL cholesterol | From baseline (week 0) to week 104
  Measured as ratio.
Change in Body Mass Index (BMI) | From baseline (week 0) to week 104
  Measured in kilograms per meter square (kg/m^2).
Number of participants who achieve BMI less than 30 kg/m^2 | At week 104
  Measured as count of participants.
Change in Glycated Haemoglobin (HbA1c) (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in HbA1c (millimoles per mole [mmol/mol]) | From baseline (week 0) to week 104
  Measured in mmol/mol.
Change in Fasting Plasma Glucose (FPG) (millimoles per liter [mmol/L]) | From baseline (week 0) to week 104
  Measured as mmol/L.
Change in FPG (milligrams per deciliter [mg/dL]) | From baseline (week 0) to week 104
  Measured as mg/dL.
Number of participants who achieve HbA1c less than (<) 5.7 percent and FPG < 100 mg/dL with prediabetes at baseline | From baseline (week 0) to week 104
  Measured as count of participants.
Number of participants who achieve HbA1c >= 6.5 percent or FPG >= 126 mg/dL with prediabetes at baseline | From baseline (week 0) to week 104
  Measured as count of participants.
Time to HbA1c < 5.7 percent and FPG < 100 mg/dL with prediabetes at baseline | From baseline (week 0) to week 104
  Measured in days.
Time to HbA1c >= 6.5 percent or FPG >= 126 mg/dL with prediabetes at baseline | From baseline (week 0) to week 104
  Measured in days.
Number of participants who develop HbA1c >= 5.7 percent or FPG greater than (>) 100 mg/dL with normoglycemia at baseline | From baseline (week 0) to week 104
  Measured as count of participants.
Number of participants who develop type 2 diabetes (T2D) as per American Diabetes Association (ADA) guideline | From baseline (week 0) to week 104
  Measured as count of participants.
Time to T2D diagnosis as per ADA guideline | From baseline (week 0) to week 104
  Measured in days.
Change in American College of Cardiology/American Heart Association (ACC/AHA) 10-year Atherosclerotic Cardiovascular Disease (ASCVD) risk score | From baseline (week 0) to week 104
  Measured in percentage of risk. American College of Cardiology/American Heart Association (ACC/AHA) risk estimator calculates 10 year risk of atherosclerotic cardiovascular disease (ASCVD) using a formula which includes age, sex, race, total cholesterol, HDL cholesterol, systolic blood pressure, blood pressure medication use, diabetes status, smoking status; minimum score 0, maximum score 100 where higher score indicates higher risk of 10-year risk of atherosclerotic cardiovascular disease (ASCVD).
Number of participants who improve in >= 1 pre-existing cardiometabolic obesity related com-plication (ORC) (hypertension, prediabetes, or dyslipidaemia) | From baseline (week 0) to week 104
  Measured as count of participants.
Ratio to baseline in C-reactive protein (CRP) | From baseline (week 0) to week 104
  Measured as ratio.
Change in total fat mass by dual energy X-ray absorption (DXA) absolute to total body mass (kilogram [kg]) | From baseline (week 0) to week 104
  Measured in kg.
Change in total fat mass by DXA relative to total body mass (kg) | From baseline (week 0) to week 104
  Measured in kg.
Change in total fat mass by DXA absolute to total body mass (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in total fat mass by DXA relative to total body mass (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in visceral fat mass by DXA, relative to baseline in visceral fat mass region (percentage) | From baseline (week 0) to week 104
  Measured in percentage.
Change in visceral fat mass by DXA, relative to total amount of fat mass in visceral fat mass region (percentage) | From baseline (week 0) to week 104
  Measured in percentage.
Change in visceral fat mass by DXA, relative to baseline in visceral fat mass region (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in visceral fat mass by DXA, relative to total amount of fat mass in visceral fat mass region (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in lean body mass by DXA absolute to total body mass (kg) | From baseline (week 0) to week 104
  Measured in kg.
Change in lean body mass by DXA relative to total body mass (kg) | From baseline (week 0) to week 104
  Measured in kg.
Change in lean body mass by DXA absolute to total body mass (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in lean body mass by DXA relative to total body mass (percentage points) | From baseline (week 0) to week 104
  Measured in percentage points.
Change in Short Form (SF)-36 Physical functioning score | From baseline (week 0) to week 104
  Measured as score points. The SF-36v2 acute measures Health-Related Quality of Life (HRQOL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. The scores are norm-based scores, i.e. transformed to a scale where the 2009 United States general population has a mean of 50 and a standard deviation of 10. Physical Functioning score ranges from 19.0-57.6, with higher scores indicating better functional health and well-being.
Change in Impact of Weight on Quality of Life-Lite for clinical trials (IWQOL-Lite-CT): Physical Function Score | From baseline (week 0) to week 104
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Physical function score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in IWQOL-Lite-CT: Physical Score | From baseline (week 0) to week 104
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Physical score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in IWQOL-Lite-CT: Psychosocial score | From baseline (week 0) to week 104
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Psychosocial score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in IWQOL-Lite-CT: Total score | From baseline (week 0) to week 104
  Measured as score points. IWQOL-Lite-CT measures weight-related physical and psychosocial functioning. The measure consists of 20 items yielding 3 composite scores, and 1 total score. Total score ranges from 0 to 100, with higher scores indicating better levels of functioning.
Change in Impact of Weight on Daily Activities Questionnaire (IWDAQ) Composite score | From baseline (week 0) to week 104
  Measured as score points. IWDAQ is an 18-item measure that uses an adaptive design to provide a personalised assessment of daily activity limitations associated with excess weight. At the baseline assessment the study participants choose the 3 activities (items) they would most like to improve the weight loss and rate the degree of limitation in each of these activities. At follow-up assessments, the study participants again rate the degree of current limitation in each of the same 3 activities. The measure yields the IWDAQ composite score with a score range from 3 to 15 with higher scores indicating greater personalised activity limitation.
Change in Control of Eating questionnaire (CoEQ): Craving Control score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional patient reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving control subscale, the subscale score is reversed so that a higher score represents a greater level of craving control.
Change in CoEQ: Positive Mood score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), and craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the Positive Mood subscale, item 6 'How anxious have you felt?' is reversed.
Change in CoEQ: Craving for Sweets score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving sweets food subscale, higher score represents a greater level of craving.
Change in CoEQ: Craving for Savoury score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving savoury food subscale, higher score represents a greater level of craving.
Change in CoEQ: Hunger score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the hunger subscale, higher score represents a greater level of craving.
Change in CoEQ: Satiety score | From baseline (week 0) to week 104
  Measured as score points. CoEQ is a 19-item multidimensional PRO that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the satiety subscale, higher score represents a greater level of craving.
CagriSema s.c. 2.4 mg/2.4 mg versus placebo: Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to week 104
  Measured as count of events.
CagriSema s.c. 2.4 mg/2.4 mg versus placebo: Number of Treatment Emergent Serious Adverse Events (TESAEs) | From baseline (week 0) to week 104
  Measured as count of events.
CagriSema s.c. 2.4 mg/2.4 mg versus CagriSema s.c. dose tapering algorithm: Number of TEAEs | From week 104 to end of study (week 162)
  Measured as count of events.
CagriSema s.c. 2.4 mg/2.4 mg versus CagriSema s.c. dose tapering algorithm: Number of TESAEs | From week 104 to end of study (week 162)
  Measured as count of events.
CagriSema 2.4 mg/2.4 mg: Number of TEAEs | From week 104 to end of study (week 162)
  Measured as count of events.
CagriSema 2.4 mg/2.4 mg: Number of TESAEs | From week 104 to end of study (week 162)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (36):
- United States (10):
  - Valley Clinical Trials, Covina, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - East West Medical Research Institute_Honolulu, Honolulu, Hawaii
  - L-MARC Research Center, Louisville, Kentucky
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group_Bristol, Bristol, Tennessee
  - North Texas Endocrine Center, Dallas, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
- Belgium (4):
  - Cliniques Universitaires Saint-Luc - Serv Endocrinologie - Diabétologie, Brussels
  - UZA - UZ Antwerpen - Department of Endocrinology, Edegem
  - UZ Leuven - Endocrinology, Leuven
  - CHU Helora - Hôpital de Mons - Site Constantinople, Mons
- Canada (4):
  - Dr. M.B. Jones Inc, Victoria, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Alpha Recherche Clinique - Lebourgneuf, Québec
- Denmark (5):
  - Aarhus Universitetshospital, Steno Diabetes Center Aarhus, Aarhus
  - Sydvestjysk Sygehus Esbjerg - Medicinsk Endokrinologisk Ambulatorium, Forskningsenheden, Esbjerg
  - Gentofte Hospital - Center for Klinisk Metabolisk Forskning, Hellerup
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
  - Sjællands Universitetshospital, Køge - Medicinsk Afdeling, Køge
- Portugal (6):
  - ULS De Matosinhos E.P.E.- Hospital Pedro Hispano, Senhora Da Hora, Matosinhos, Matosinhos
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - CUF Descobertas, Lisbon
  - Hospital Cuf Descobertas S.A., Lisbon
  - Unidade Local de Saude de Sao Joao E.P.E, Porto
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
- United Kingdom (7):
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital_Cambridge, Cambridge
  - University Hospital Coventry - WISDEM Centre, Coventry
  - Aintree University Hospital, Liverpool
  - Royal London Hospital - Blizard Institute, London
  - Joint Clinical Research Facility - Swansea, Swansea
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com